CLINICAL TRIAL: NCT00102401
Title: Comparing the Effects of an Internet-Based to an Established Dyspnea Self-Management Program on Dyspnea, Exercise Behavior, and Pulmonary Exacerbations in Patients With COPD
Brief Title: Internet-Based and Established Dyspnea Self-Management Programs in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49153
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Pulmonary Disease, chronic obstructive; Lung disease, obstructive; Self-care; Self-management; Patient education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive

INTERVENTIONS:
Behavioral: Internet-based Dyspnea Self-Management Program
Behavioral: Face-to-face Dyspnea Self-Management Program

SUMMARY:
The overall goal of this study is to compare the impact of a new Internet Dyspnea Self-Management Program (eDSMP) with an established face-to-face Dyspnea Self-Management Program (DSMP) in patients with COPD. The primary aim of the study is to test the following two hypotheses: 1. The eDSMP and the DSMP will have comparable improvements in the primary outcomes of shortness of breath (dyspnea) with activities of daily living (ADL), exercise adherence and performance, and pulmonary exacerbations (frequency and duration) at 3 and 6 months. 2. The eDSMP and the DSMP will have comparable improvements in the secondary outcomes of perception of support, self-efficacy for exercise and managing dyspnea, and health resource utilization at 3 and 6 months. This study is a randomized, longitudinal, repeated measures design with measurement times at 0, 3, and 6 months.

DETAILED DESCRIPTION:
Despite optimal medical treatment, people with chronic obstructive pulmonary disease (COPD) continue to experience dyspnea or shortness of breath. This study will evaluate two different ways to provide education and support to help patients manage their shortness of breath. One program will be conducted in a face-to-face setting and a second through the Internet. The main difference between the two programs is the way they are administered. The education, exercise, and monitoring components are the same. The overall goal of this study is to find out whether the two programs are comparable in their effect on shortness of breath (dyspnea) with activities of daily living, exercise adherence and performance, and pulmonary exacerbations (frequency and duration) at 3 and 6 months. Perception of support, self-efficacy for exercise and managing dyspnea, and health resource utilization will also be measured at 3 and 6 months. This study is a randomized, longitudinal, repeated measures design with measurement times at 0, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD, clinically stable for 1 month;
* Spirometry results showing at least mild disease (FEV1/FVC < 70% and FEV1 < 80% predicted after bronchodilator);
* ADL limited by dyspnea;
* Ability to speak English and sign consent form;
* Actively use computer and the Internet;
* Maintain O2 saturation > 85% on < 6 L/min of nasal oxygen during the six minute walk;
* Understands and is able to rate shortness of breath during exercise

Exclusion Criteria:

* Active symptomatic illness other than COPD;
* Formal pulmonary rehabilitation training in the past 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Dyspnea
Exercise adherence and performance
Pulmonary exacerbations

SECONDARY OUTCOMES:
Perception of support
Self-efficacy for exercise and managing dyspnea
Health resource utilization

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Carrieri-Kohlman, RN DNSc, Principal Investigator — University of California, San Francisco; Huong Q Nguyen, RN PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - University of California, San Francisco, California
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Fu H, Garrett B, Tao G, Cordingley E, Ofoghi Z, Taverner T, Sun C, Cheung T. Virtual Reality-Guided Meditation for Chronic Pain in Patients With Cancer: Exploratory Analysis of Electroencephalograph Activity. JMIR Biomed Eng. 2021 Jun 24;6(2):e26332. doi: 10.2196/26332. PMID 38907380
- [Derived] Chung A, Seixas A, Williams N, Senathirajah Y, Robbins R, Newsome Garcia V, Ravenell J, Jean-Louis G. Development of "Advancing People of Color in Clinical Trials Now!": Web-Based Randomized Controlled Trial Protocol. JMIR Res Protoc. 2020 Jul 14;9(7):e17589. doi: 10.2196/17589. PMID 32673274
- [Derived] Greysen SR, Magan Y, Rosenthal J, Jacolbia R, Auerbach AD, Harrison JD. Patient Recommendations to Improve the Implementation of and Engagement With Portals in Acute Care: Hospital-Based Qualitative Study. J Med Internet Res. 2020 Jan 14;22(1):e13337. doi: 10.2196/13337. PMID 31934868
- [Derived] Arostegui I, Legarreta MJ, Barrio I, Esteban C, Garcia-Gutierrez S, Aguirre U, Quintana JM; IRYSS-COPD Group. A Computer Application to Predict Adverse Events in the Short-Term Evolution of Patients With Exacerbation of Chronic Obstructive Pulmonary Disease. JMIR Med Inform. 2019 Apr 17;7(2):e10773. doi: 10.2196/10773. PMID 30994471
- [Derived] Abbott-Garner P, Richardson J, Jones RB. The Impact of Superfast Broadband, Tailored Booklets for Households, and Discussions With General Practitioners on Personal Electronic Health Readiness: Cluster Factorial Quasi-Randomized Control Trial. J Med Internet Res. 2019 Mar 11;21(3):e11386. doi: 10.2196/11386. PMID 30855234
- [Derived] McHugh J, Lee O, Aspell N, Lawlor BA, Brennan S. A shared mealtime approach to improving social and nutritional functioning among older adults living alone: study protocol for a randomized controlled trial. JMIR Res Protoc. 2015 Apr 21;4(2):e43. doi: 10.2196/resprot.4050. PMID 25900904
- [Derived] Nguyen HQ, Donesky-Cuenco D, Wolpin S, Reinke LF, Benditt JO, Paul SM, Carrieri-Kohlman V. Randomized controlled trial of an internet-based versus face-to-face dyspnea self-management program for patients with chronic obstructive pulmonary disease: pilot study. J Med Internet Res. 2008 Apr 16;10(2):e9. doi: 10.2196/jmir.990. PMID 18417444